CLINICAL TRIAL: NCT00023400
Title: TBTC Study 23B:Intensive Pharmacokinetics of the Nelfinavir Rifabutin Interaction in Patients With HIV-Related Tuberculosis Treated With a Rifabutin-Based Regimen
Brief Title: TBTC Study 23B:Intensive PK of the Nelfinavir Rifabutin Interaction in Patients With HIV-TB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-2587; 23B
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections; Tuberculosis
Keywords: tuberculosis; TB
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Nelfinavir; Rifabutin

INTERVENTIONS:
Drug: Nelfinavir
Drug: Rifabutin

SUMMARY:
Primary Objective:

To define the impact of nelfinavir (given at 1250mg bid as part of a combination antiretroviral regimen) on peak levels and area under the curve for rifabutin and the rifabutin metabolite, 25-O-desacetyl rifabutin when rifabutin is given at 300 mg bi-weekly as part of tuberculosis chemotherapy.

Secondary Objectives:

To compare the pharmacokinetics of nelfinavir given twice daily at 1250 mg bid with twice-weekly isoniazid and rifabutin to the pharmacokinetics of nelfinavir 1250 mg twice-daily in historical HIV-infected patients not receiving isoniazid and rifabutin.

To evaluate the correlation between pharmacokinetic parameters of rifabutin and 25-O-desacetyl rifabutin and the occurrence of toxicity attributed to rifabutin in patients with HIV-related tuberculosis.

To define detailed pharmacokinetics of isoniazid given at 15mg/kg or 900 mg in patients with HIV-related tuberculosis.

To attempt to derive optimal sampling times for nelfinavir and rifabutin pharmacokinetic studies.

ELIGIBILITY:
* Patients with HIV-related tuberculosis

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2000-02; Study Completion 2002-02

PRIMARY OUTCOMES:
Impact of nelfinavir (given at 1250mg bid as part of a combination antiretroviral regimen) on area under the curve for rifabutin and 25-O-desacetyl rifabutin when rifabutin is given 300 mg bi-weekly as part of tuberculosis chemotherapy.

SECONDARY OUTCOMES:
To compare the pharmacokinetics of nelfinavir given twice daily at 1250 mg bid with twice-weekly isoniazid and rifabutin to the pharmacokinetics of nelfinavir 1250 mg twice-daily in historical HIV-infected patients not receiving isoniazid and rifabutin.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Benator, MD, Study Chair — Washington, D.C. VAMC
Locations (23):
- United States (20):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Washington, D.C. VAMC, Washington D.C., District of Columbia
  - Chicago VA Medical Center (Lakeside), Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New Jersey Medical School, Newark, New Jersey
  - New York University School of Medicine, New York, New York
  - Columbia University/Presbyterian Medical Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nashville VA Medical Center, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Thomas Street Clinic, Houston, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Montreal Chest Institute McGill University, Montreal, Quebec

REFERENCES:
- See also: (Click here for more information about the Tuberculosis Trials Consortium(TBTC) — http://www.cdc.gov/nchstp/tb/tbtc/